CLINICAL TRIAL: NCT00508430
Title: ASP 8825 Phase II Study-A Double- Blind, Placebo- Controlled Study in Patients With Painful Diabetic Polyneuropathy
Brief Title: ASP 8825 - Study in Patients With Painful Diabetic Polyneuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: An independent DMC determined continuation was unlikely to demonstrate a statistically significant advantage of ASP8825 over placebo on the primary endpoint
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8825-CL-0007
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-12

CONDITIONS: Diabetic Neuropathies
Keywords: ASP8825; Diabetic Neuropathies; Pain
MeSH Terms: conditions — Diabetic Neuropathies; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Low dose group
  Interventions: Drug: ASP8825
- 2 (Experimental): Middle dose group
  Interventions: Drug: ASP8825
- 3 (Experimental): High dose group
  Interventions: Drug: ASP8825
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP8825 — oral
  Arms: 1; 2; 3
Drug: Placebo — oral
  Arms: 4

SUMMARY:
To demonstrate the superiority of ASP8825 over placebo and dose response in patients with painful diabetic polyneuropathy.

DETAILED DESCRIPTION:
Three doses of ASP8825 are compared to placebo in efficacy and safety point of view in patients with painful diabetic polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 20 - 79 years
* Diabetes mellitus patients with diabetic polyneuropathy who have pain symptom for 26 weeks prior to the study
* Subjects who are compliant with diary completion

Exclusion Criteria:

* Subjects who have pain from other diseases at the evaluating site
* Subjects who have nerve diseases at the evaluating site
* Subjects with foot ulcer or gangrene

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2007-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Pain severity rating | 8 week

SECONDARY OUTCOMES:
Severity of numbness, maximum pain, night pain and sleep disturbance. | 8 week
Responder rate | 8 week
Patient's global impression of change | 8 week
Clinical's global impression of change | 8 week

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kanto
  - Kyusyu
  - Shikoku
  - Tōhoku